CLINICAL TRIAL: NCT06752811
Title: A Multi-center, Randomized, Open, Parallel-group, Positive Drug-controlled Phase III Clinical Trial for Evaluating the Efficacy and Safety of Paclitaxel Polymeric Micelles for Injection Plus Gemcitabine and Paclitaxel for Injection (Albumin-bound) Plus Gemcitabine for Injection in the First-line Treatment of Metastatic Pancreatic Cancer
Brief Title: Polymeric Micellar Paclitaxel for Metastatic Pancreatic Cancer
Acronym: pompom
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Yizhong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai Yizhong
Record Dates: First submitted 2024-12-20; First posted 2024-12-31 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer Metastatic
Keywords: paclitaxel polymeric micelles for injection
MeSH Terms: interventions — Injections; Gemcitabine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- paclitaxel polymeric micelles for injection+Gemcitabine Hydrochloride for Injection (Experimental): Patients in the experimental group will receive intravenous infusion of paclitaxel polymeric micelles for injection at a dose of 300 mg/m2 (based on body surface area), administered on Day 1, with intravenous infusion for ≥ 3 hours, every 3 weeks as a cycle. Then, the subjects also need to receive intravenous infusion of gemcitabine hydrochloride combination therapy at a dose of 1000 mg/m2 (based on body surface area), administered at D1 and D8 every 3 weeks.
  Interventions: Drug: paclitaxel polymeric micelles for injection; Drug: Gemcitabine Hydrochloride for Injection
- paclitaxel for injection(albumin bound )+Gemcitabine Hydrochloride for Injection (Active Comparator): Control Group: Patients in the control group will receive intravenous infusion of paclitaxel (albumin bound) at a dose of 125 mg/m2 (based on body surface area), administered at D1, D8, and D15, every 4 weeks as a cycle. Then, the subjects also need to receive intravenous infusion of gemcitabine hydrochloride combination therapy at a dose of 1000 mg/m2 (based on body surface area), administered at D1, D8, and D15 every 4 weeks.
  Interventions: Drug: Paclitaxel for Injection (albumin bound ); Drug: Gemcitabine Hydrochloride for Injection

INTERVENTIONS:
Drug: paclitaxel polymeric micelles for injection — Paclitaxel polymeric micelles for injection at a dose of 300 mg/m2 (based on body surface area), administered on Day 1, with intravenous infusion for ≥ 3 hours, every 3 weeks as a cycle.
  Arms: paclitaxel polymeric micelles for injection+Gemcitabine Hydrochloride for Injection
Drug: Gemcitabine Hydrochloride for Injection — The subjects also need to receive intravenous infusion of gemcitabine hydrochloride combination therapy at a dose of 1000 mg/m2 (based on body surface area), administered at D1 and D8 every 3 weeks.
  Arms: paclitaxel polymeric micelles for injection+Gemcitabine Hydrochloride for Injection
Drug: Paclitaxel for Injection (albumin bound ) — Patients in the control group will receive intravenous infusion of paclitaxel for Injection (albumin bound ) at a dose of 125 mg/m2 (based on body surface area), administered at D1, D8, and D15, every 4 weeks as a cycle.
  Arms: paclitaxel for injection(albumin bound )+Gemcitabine Hydrochloride for Injection
Drug: Gemcitabine Hydrochloride for Injection — The subjects also need to receive intravenous infusion of gemcitabine hydrochloride combination therapy at a dose of 1000 mg/m2 (based on body surface area), administered at D1, D8, and D15 every 4 weeks.
  Arms: paclitaxel for injection(albumin bound )+Gemcitabine Hydrochloride for Injection

SUMMARY:
This trial is a multi-center, randomized, open, parallel-group and positive-controlled phase III trial to evaluate the efficacy and safety of paclitaxel polymeric micelles for injection plus gemcitabine as first-line treatment of metastatic pancreatic cancer compared with nab-Paclitaxel plus gemcitabine.

DETAILED DESCRIPTION:
Based on the widespread use of paclitaxel in pancreatic cancer, this study aims to develop a clinical protocol of paclitaxel polymeric micelles for injection in combination with gemcitabine as first-line treatment for metastatic pancreatic cancer, in order to find a more effective treatment option for pancreatic patients and thus improve survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1) Men or women aged 18 to 75 years old (including the critical value).
* 2）Metastatic pancreatic cancer confirmed by histology or cytology.
* 3）Patients who have not previously received any systemic therapy (including chemotherapy, targeted, and immunotherapy), radiotherapy, surgery, or investigational drugs for the treatment of metastatic pancreatic cancer; Patients who have previously received neoadjuvant or adjuvant chemotherapy could be enrolled if the interval between last treatment and recurrence and metastasis is more than 6 months.
* 4）Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* 5）Survival is expected to be at least 3 months.
* 6）At least one metastatic lesion (non-lymph node lesions with a major diameter of ≥ 10 mm on CT or MRI and lymph node lesions with a minor diameter of ≥ 15 mm) that is measurable according to the Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) and is amenable to accurate repeated measurement. Suspected metastatic lesions (non-regional lymph nodes) that do not meet the above measurable standards and the primary lesions are measurable, the metastatic lesions are confirmed pathologically, can also be included.
* 7）The major organs function well: a) white blood cell count ≥ 3.0 × 10^9/L. b) Hemoglobin ≥ 90.0 g/L. c) Absolute neutrophil count ≥1.5 × 10^9/L. d) Platelet count ≥100 × 10^9/L. e) Total bilirubin ≤1.5 × upper limit of normal range (ULN). f) Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 2.5 × ULN; For patients with liver metastasis, ALT, AST and ALP ≤ 5 × ULN; ALP ≤ 10 × ULN in patients with bone metastases.

  g) Serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance estimated by Cockcroft Gault formula ≥50 ml/min.

  h) International normalized ratio (INR) ≤ 1.5 × ULN and prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
* 8）Women of childbearing age are required to have a negative pregnancy test at the screening period and to use a highly effective contraceptive method for 6 months from the screening period to the last dose. Male participants whose partners are women of childbearing age are required to use a highly effective contraceptive method for 6 months after the first dose of a trial product until the last dose.
* 9）Patients are able to understand the steps of this trial, are willing to follow the clinical trial protocol to complete the trial, and sign the Informed Consent Form.

Exclusion Criteria:

* 1）Patients who are allergic to the investigational drugs and their analogues, or excipients.
* 2）Patients who had any other malignant tumors within 5 years before or at present, except those who had been completely cured, such as basal cell carcinoma, skin squamous cell carcinoma, melanoma in situ, papillary thyroid carcinoma and cervical carcinoma in situ, were excluded.
* 3）CNS (central nervous system) or meningeal metastases are known, except for those with single brain metastases that are strictly controlled and asymptomatic.
* 4）Patients with tumor liver metastasis exceeding 1/2 of the entire liver during screening; or there may be active hepatitis B (HBsAg test positive, HBV-DNA>500 IU/ml or research center detection limit [only when the research center limit is above 500 IU/ml]); Active hepatitis C (positive for hepatitis C virus (HCV) antibodies and HCV-RNA > research center detection limit).
* 5） Human Immunodeficiency Virus test is positive.
* 6）Patients with active, uncontrolled bacterial, viral, or fungal infection requiring current systemic anti-infective therapy.
* 7） Patients who have a history of drug or alcohol abuse prior to screening.
* 8）Patients with severe organic lesions or major organ failure, such as decompensated heart and lung failure, leading to intolerance to chemotherapy.
* 9） Patients with bleeding tendency (e.g., presence of active ulcer lesions in stomach, melena and/or hematemesis within 3 months, hemoptysis).
* 10） History of severe cardiovascular and cerebrovascular diseases, including but not limited to:

  1. NYHA (New York Heart Association) class III or IV heart disease;
  2. Uncontrollable hypertension (i.e. systolic blood pressure ≥ 160 mmHg, and/or diastolic blood pressure ≥ 100 mmHg)；
  3. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, II-III degree atrioventricular block, etc;
  4. QT interval prolongation corrected for heart rate (corrected for QTc interval using Fridericia formula, males>450ms, females>470ms);
  5. Individuals with significant abnormalities in electrocardiogram with clinical significance;
  6. Acute coronary syndrome, congestive heart failure, stroke, or other grade 3 or higher cardiovascular events occurring within 6 months prior to the first administration;
* 11） Clinically uncontrollable third space effusion, such as pleural effusion, pericardial effusion, peritoneal effusion, etc. If there were no clinical symptoms, small amounts of pleural effusion or ascites that did not require clinical intervention could be enrolled only after strict control.
* 12） serious psychiatric disorders in the past or current.
* 13）Organ transplant recipients.
* 14）Use of the prohibited medications specified in the protocol is planned during the screening and treatment periods.
* 15） Patients with a history of psychotropic drug abuse and unable to quit.
* 16）Before screening, participants have participated in another clinical trial with an investigational nonbiologic agent (administered within the past 30 days or five half-lives, whichever was longer) or an investigational biologic agent (monoclonal or polyclonal antibody) (within the past 4 months or five half-lives, whichever is longer).
* 17）Pregnant or lactating female patients.
* 18）Participants who are judged by the investigator to be unable to follow trial procedures or who are judged by the investigator to be unfit to participate in the trial for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | Randomization to measured PD or date of death from any cause（up to 36 months)
  PFS(Progression-Free-Survival) is the time from randomization until the date of objectively determined progressive disease (PD) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival(OS) | Randomization to date of death from any cause（up to 36 months)
  The time from randomization to death.
Objective Response Rate(ORR) | Baseline to measured PD（up to 36 months)
  Proportion of subjects who have achieved complete response (CR) or partial response (PR) (RECIST 1.1)
Disease Control Rate（DCR） | Baseline to measured PD（up to 36 months)
  Proportion of subjects who have achieved complete response (CR), partial response (PR) or stable disease (SD) (RECIST 1.1)
Incidence of adverse events | up to 36 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0".

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No